CLINICAL TRIAL: NCT05447871
Title: Single-injection Modified 4 in 1 Block Versus Adductor Canal Block as Postoperative Analgesia in Total Knee Arthroplasty
Brief Title: Single-injection Modified 4 in 1 Block as Postoperative Analgesia in Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MFM-IRB: MD. 22.03.629
Record Dates: First submitted 2022-06-22; First posted 2022-07-07 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Total Knee Arthroplasty

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single blind (participant) study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound guided single injection modified 4 in 1 block technique (Experimental): Patients in this group will receive ultrasound guided single injection modified 4 in 1 block with 25 ml bupivacaine 0.25%
  Interventions: Procedure: Ultrasound guided single injection modified 4 in 1 block technique; Drug: Bupivacaine 0.25%
- Ultrasound guided adductor canal block technique (Active Comparator): Patients in this group will receive ultrasound guided aduuctor canal block with 20 ml bupivacaine 0.25%
  Interventions: Procedure: Ultrasound guided adductor canal block technique; Drug: Bupivacaine 0.25%

INTERVENTIONS:
Procedure: Ultrasound guided single injection modified 4 in 1 block technique — A high-frequency ultrasound probe is placed over the femoral condyle and vastus medialis muscle is identified. The probe is slid proximally till the superficial femoral artery appeared. The probe is slid proximally till the descending genicular artery branching from the superficial femoral artery. The point of interest is 8-10 cm above the femoral condyle. The needle is guided into the Vastus medialis muscle till the nerve to Vastus medialis. At this point, 5-7 mL of the local anaesthetic drug is injected. The needle is guided further in-plane from lateral to medial side to reach the perivascular region and after negative aspiration 25 ml local anaesthetic drug is injected.
  Arms: Ultrasound guided single injection modified 4 in 1 block technique
Procedure: Ultrasound guided adductor canal block technique — The Adductor canal is identified in the middle of the thigh beneath the sartorius muscle using a high-frequency ultrasonic transducer. the probe is slid till the superficial femoral artery appeared in the adductor canal between vastus medialis and adductor longus muscle. A 22-gauge spinal needle is inserted in a lateral to medial plane to reach the perivascular region and after negative aspiration 20 ml local anaesthetic drug is injected, visualised to push the femoral artery.
  Arms: Ultrasound guided adductor canal block technique
Drug: Bupivacaine 0.25% — bupivacaine 0.25%

SUMMARY:
Patients suffer from moderate to severe pain after TKA. Patients are asked to begin functional exercise as early as possible after surgery, and that requires adequate control of postoperative pain. Regional anesthesia divides into non-motor sparing peripheral nerve blocks as femoral n. block and sciatic n. block and motor sparing peripheral nerve block as adductor canal block and IPACK but these blocks have many drawbacks.

So new studies found that a modified 4 in-1 block blocks all these nerves and produces adequate analgesia without sparing areas.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) is regarded as the most effective method to reduce knee pain and improve knee function in patients with advanced knee osteoarthritis. Postoperative pain is an unpleasant experience for TKA and this pain might greatly influence patients' early rehabilitation.

Almost 60% of patients suffer moderate to severe pain after TKA and 25% of them could even develop related complications, such as longer hospitalization stays, unanticipated hospital admissions, readmissions, etc.

With the development of enhanced recovery after surgery, patients are asked to begin exercise as early as possible after surgery, and that requires adequate control of postoperative pain.

Multimodal systemic analgesia plays an essential role in controlling postoperative pain after TKA by controlling the inflammatory process, dealing with the neuropathic component of pain, and thus reducing the severity of pain.

Multimodal analgesia includes more than one pain-control modality (systemic analgesia and regional anaesthesia). Systemic analgesia includes acetaminophen, nonsteroidal anti-inflammatory drugs, steroids and opioids. Regional anaesthesia includes epidural analgesia, femoral n. block, adductor canal block, sciatic n. block, IPACK, etc. Regional anaesthesia divides into non-motor sparing peripheral nerve blocks as femoral n. block and sciatic n. block and motor sparing peripheral nerve block as adductor canal block and IPACK.

But these blocks have many drawbacks. Femoral n. block is associated with quadriceps muscle weakness leading to delay in patient's mobility. Sciatic n. block also causes foot drop. The Adductor canal block does not cover the skin on the back of the knee. Surgeons refuse IPACK because of diffusion of local anaesthetics disturbs the anatomy of the surgical field.

The Modified 4 in 1 block technique aims to block four nerves (saphenous nerve, obturator nerve, nerve to vastus medialis and sciatic nerve) through a single injection point by spreading up to the adductor canal in midthigh and below to the popliteal fossa. The investigator will conduct this randomized clinical trial to evaluate the quality of postoperative analgesia produced by a single injection modified 4 in 1 block and midsartorius adductor canal block with regard to total analgesic consumption in the first 24 hours postoperatively

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) of 19-30 kg/m2
* American Society of Anesthesiologists (ASA) functional status of I-III

Exclusion Criteria:

* Drug hypersensitivity
* coagulopathy
* infection at the site of injection
* Traumatic arthirits

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Total amount of postoperative analgesia in first 24 hours | in first 24 hours
  calculate total amount of morphine hydrochloride which patient will need in first 24 hours postoperative.

SECONDARY OUTCOMES:
Duration of sensory block. | 3, 6, 12, 24 hours postoperative
  return of pinbrick sensation on the lateral aspect of the foot (S1)
Duration of motor block. | 3, 6, 12, 24 hours postoperative
  motor block is tested and recoded every 30 min till Bromage score is zero
Total distance patient will be able to ambulate on first postoperative day | on first postoperative day
  the distance that patient will be able to walk on the first postoperative day (meters)
intraoperative non invasive blood pressure(NIBP) mmHg | every 10 minutes after spinal anesthesia till the end of the surgery
  NIBP will be measured and recorded.
intraoperative heart rate beat per minute | every 10 minutes after spinal anesthesia till the end of the surgery.
  heart rate will be monitored and recorded.
postoperative hypotension mmHg | at 1, 3, 6, 12 hours postoperative
  blood pressure will be measured and recorded

CONTACTS AND LOCATIONS:
Overall Officials: Gehan A Trabeeh, MD, Study Chair — Professor of Anesthesia and Surgical Intensive Care; Samah A Gouda, MD, Study Director — Assistant Professor of Anesthesia and Surgical Intensive Care; Samar A Alattar, M.Sec, Principal Investigator — Assistant lecturer of Anesthesia and Surgical Intensive Care
Locations (1):
- Mansoura University, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Yes, Study Protocol Statistical Analysis Plan (SAP) Informed Consent Form (ICF) Clinical Study Report (CSR) Supporting Information:
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: after completing the study and being accepted for publication.After six months after completing the study.
Access Criteria: The data will be accessible to the investigators and PRS administrators with hiding the identifiers for the patients.